CLINICAL TRIAL: NCT06850441
Title: Effects of Anti-Stigma Psychoeducation Based on Roy Adaptation Model on Stigma and Quality of Life in Individuals With Type 1 Diabetes
Brief Title: Effects of Education on Stigma and Quality of Life in Individuals With Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ece MUTLU SATIL, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IzmirKCU-SBF-EMS-001
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type I; Stigma; Quality of Life (QOL)
Keywords: Diabetes Mellitus, Type I; Stigma; Quality of life; Roy Adaptation Model
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Social Stigma

STUDY DESIGN:
Intervention Model Description: Intervention group to be given group psychoeducation The control group to continue their routine treatments and not receive intervention
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A diabetes education nurse will identify participants and assign numbers to the identified participants. A statistician will randomize the participant numbers. A different nurse will place the participants in the experimental and control groups according to the numbers.
  A statistician will evaluate the results of the education. Thus, the researcher will be blinded in both the participant selection and the outcome evaluation stages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Group (Experimental): The education is a group psychoeducation. Education methods such as role-play, discussion, demonstration, and narration will be applied. The education will be held once a week and will be completed in 7 weeks.
  Psychoeducation topics include adaptation to stigma in type 1 diabetes, coping, diabetes management, social life, self-esteem, roles in life and impact on life. Concepts such as stigma, blame, judgment, discrimination, shame and stereotyped thoughts will be included.
  Interventions: Other: Psychoeducation
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Psychoeducation — The education is a group psychoeducation. Education methods such as role-play, discussion, demonstration, and narration will be applied. The education will be held once a week and will be completed in 7 weeks.
  Psychoeducation topics include adaptation to stigma in type 1 diabetes, coping, diabetes management, social life, self-esteem, roles in life and impact on life. Concepts such as stigma, blame, judgment, discrimination, shame and stereotyped thoughts will be included.
  Arms: Psychoeducation Group

SUMMARY:
This clinical trial aimed to examine the effects of anti-stigma psychoeducation based on the Roy Adaptation Model on stigma and quality of life in individuals with Type 1 Diabetes.The main questions it aims to answer are:

1. Does anti-stigma psychoeducation reduce stigma of individuals diagnosed with Type 1 Diabetes?
2. Does anti-stigma psychoeducation improve the quality of life of individuals diagnosed with Type 1 Diabetes?

Researchers will compare the group that did not receive stigma prevention psychoeducation with those that did.

Participants will receive 7 sessions of the psychoeducation once a week. An evaluation session will be administered 3 months after the psychoeducation.

Researchers will assess all participants' stigma and quality of life before, after and 3 months after the psychoeducation.

DETAILED DESCRIPTION:
Individuals who were diagnosed with Type 1 Diabetes at least 6 months ago, are between the ages of 18-75, and can speak and understand the language spoken will be included in the study. Individuals with hearing and visual impairments and those diagnosed with mental retardation will not be included in the study. Participants will be assigned to the intervention and control groups by the statistician through randomization. Each group will consist of 18 people.

Stigma prevention psychoeducation will be applied to the intervention group. This psychoeducation will be conducted as a group education. No intervention will be applied to the control group.

The researcher will evaluate the stigma and quality of life of the intervention and control groups before, after and 3 months after the education. pre-test and post-test and 3-month follow-up Group psychoeducation will be applied to the participants in the intervention group once a week. After the education, they will be evaluated according to the nursing outcome criteria

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 diabetes at least 6 months ago,
* Being between the ages of 18 and 75,
* Speaking and understanding Turkish,

Exclusion Criteria:

* Having hearing and vision impairment
* Being diagnosed with mental retardation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Type 1 Diabetes Stigma Assessment Scale | 0 day, 7 weeks, 3 months
  Type 1 Diabetes Stigma Assessment Scale was developed by Browne et al. in 2017 to assess perceived and experienced stigma in adults diagnosed with type 1 diabetes. The scale consists of 19 items. The scale has 3 sub-dimensions; "treated differently", "Blame and judgment" and "Identity concerns" Each item is scored on a 5-point Likert scale. (1=strongly disagree, 2=disagree, 3=not sure, 4=agree, 5=strongly agree). Item scores are added to obtain the sub-dimensions and total score of the scale. A high score indicates an increase in perceived and felt stigma.

SECONDARY OUTCOMES:
Short Form-36 | 0 day, 7 weeks, 3 months
  Short Form-36 is a scale that evaluates quality of life in terms of physical and mental health. It was developed by Ware and his colleagues (Ware and Sherbourne, 1992). It consists of 36 items and 8 sub-dimensions; Physical function, physical role, pain, general health perception, vitality, social function, mental role and mental health. The 4th and 5th items of the assessment are yes/no and the rest are Likert type. The sub-dimensions are scored, not the whole scale. The scoring of the sub-scales varies between 0 and 100. A high score indicates a better level of health, while a low score indicates deterioration in health.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Dülgerler, PhD, Study Chair — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This experimental study is a thesis study. In order to preserve originality, I do not approve of sharing it.

REFERENCES:
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Browne JL, Ventura AD, Mosely K, Speight J. Measuring Type 1 diabetes stigma: development and validation of the Type 1 Diabetes Stigma Assessment Scale (DSAS-1). Diabet Med. 2017 Dec;34(12):1773-1782. doi: 10.1111/dme.13507. PMID 28891210
- [Result] Satil EM, Arabaci LB. Turkish validity and reliability of Type-1 Diabetes Stigma Assessment Scale. North Clin Istanb. 2022 Dec 12;9(6):654-662. doi: 10.14744/nci.2021.36937. eCollection 2022. PMID 36685628